CLINICAL TRIAL: NCT02834715
Title: Effects of Stevia on Glycaemic Profile and Insulin Secretion of Type 2 Diabetic Patients
Brief Title: Metabolic Effects of Stevia in Type 2 Diabetic Patients
Acronym: STEDIA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor, Yaounde Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNO20161
Record Dates: First submitted 2016-07-08; First posted 2016-07-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Stevia; insulin secretion; insulin sensitivity; Sweetener
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stevia (Experimental): Once-daily oral intake of 240 mg of Stevia liquid extract for 30 days as food supplement.
  Interventions: Dietary Supplement: Stevia rebaudiana liquid extract
- Control (No Intervention): No intervention, similar follow up as experimental arm to control for trial effect

INTERVENTIONS:
Dietary Supplement: Stevia rebaudiana liquid extract — Sweetener made of liquid stevia self administered daily for 30 days
  Arms: Stevia

SUMMARY:
The main aim of the study is to assess the short term and 1-month metabolic effects of Stevia rebaudiana bertoni in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This is a non-randomized clinical trial in a type 2 diabetic population aiming to investigate the effect of Stevia rebaudiana bertoni on the glycaemic and insulin secretory response to a mixed meal tolerance test, insulin sensitivity and lipid profile. The study has two arms including an intervention arm (test group) and a non-intervention arm (controls) matched for age, sex and body mass index in 2:1 ratio.

The intervention is made of two phases including

1. A mixed meal tolerance test with and without 240 mg of Stevia in a randomized order to evaluate the acute effects;
2. An oral intake of 240 mg of Stevia within 30 days as food supplement in order to assess medium-term effects

ELIGIBILITY:
Inclusion Criteria:

* Known type 2 diabetes
* Unchanged hypoglycaemic treatment for at least 3 months prior to inclusion
* No acute complication of diabetes
* HbA1C≤ 8%

Exclusion Criteria:

* Infection up to 10 days prior to inclusion
* Serum ALAT >3N,
* MDRD estimated creatinine clearance <60ml/min
* Tobacco smoking

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Glycaemic profile in response to mixed meal test | 1 month
  Change in blood glucose profile during a mixed meal test at baseline and after one month intervention

SECONDARY OUTCOMES:
insulin secretion in response to mixed meal test | 1 month
  Change in serum C-peptide profile during a mixed meal test at baseline and after one month intervention
Serum lipids | 1 month
  Change in fasting serum lipids
Insulin sensitivity | 1 month
  Change in mixed meal derived insulin sensitivity
Liver enzymes | 1 month
  Change in serum alanine amino transferase

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sobngwi, MD, PhD, Principal Investigator — University of Yaoundé 1 and Yaoundé Central Hospital
Locations (1):
- National Obesity Centre, Yaoundé, Cameroon